CLINICAL TRIAL: NCT02311361
Title: A Pilot Study of Immune Checkpoint Inhibition (Durvalumab With or Without Tremelimumab) in Combination With Radiation Therapy in Patients With Unresectable Pancreatic Cancer
Brief Title: Immune Checkpoint Inhibition (Tremelimumab and/or MEDI4736) in Combination With Radiation Therapy in Patients With Unresectable Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Tim Greten, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 150027; 15-C-0027
Record Dates: First submitted 2014-12-05; First posted 2014-12-08 (Estimated); Results first posted 2020-07-17 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-03

CONDITIONS: Pancreatic Neoplasms; Pancreatic Cancer; Cancer of Pancreas; Cancer of the Pancreas; Pancreas Cancer
Keywords: Anti-PDL1; Anti-CTLA4; Streostatic Body Radiation Therapy (SBRT); Monoclonal Antibody; Antitumor Immunity
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Durvalumab + 8 Gray (Gy) in 1 fraction (Experimental): Cohort 1/Dose Level A1 Durvalumab + 8 Gray (Gy) in 1 fraction
  Interventions: Biological: Durvalumab; Radiation: Sterostatic body radiation therapy (SBRT)
- Durvalumab +5 Gy in 5 fractions (Experimental): Cohort 2/Dose Level A2 Durvalumab +5 Gy in 5 fractions
  Interventions: Biological: Durvalumab; Radiation: Sterostatic body radiation therapy (SBRT)
- Tremelimumab + 8 Gy in 1 fraction (Experimental): Cohort 3/Dose Level B1 (was removed with Amendment A) Tremelimumab + 8 Gy in 1 fraction
  Interventions: Biological: Tremelimumab; Radiation: Sterostatic body radiation therapy (SBRT)
- Tremelimumab + 5 Gy in 5 fractions (Experimental): Cohort 4/Dose Level B2 (was removed with Amendment A) Tremelimumab + 5 Gy in 5 fractions
  Interventions: Biological: Tremelimumab; Radiation: Sterostatic body radiation therapy (SBRT)
- Durvalumab +Tremelimumab + 8 Gy in 1 fraction (Experimental): Cohort C/ Dose Level C1 Durvalumab +Tremelimumab + 8 Gy in 1 fraction
  Interventions: Biological: Durvalumab; Biological: Tremelimumab; Radiation: Sterostatic body radiation therapy (SBRT)
- Durvalumab +Tremelimumab +5 Gy in 5 fractions (Experimental): Cohort C/Dose Level C2 Durvalumab +Tremelimumab +5 Gy in 5 fractions
  Interventions: Biological: Durvalumab; Biological: Tremelimumab; Radiation: Sterostatic body radiation therapy (SBRT)

INTERVENTIONS:
Biological: Durvalumab — 10 mg/kg, mg intravenous (IV), every two weeks, or 1500 mg, IV, every four weeks.
  Other Names: MEDI4736
  Arms: Durvalumab + 8 Gray (Gy) in 1 fraction; Durvalumab +5 Gy in 5 fractions; Durvalumab +Tremelimumab + 8 Gy in 1 fraction; Durvalumab +Tremelimumab +5 Gy in 5 fractions
Biological: Tremelimumab — 75 mg IV, every 4 weeks for 16 weeks
  Other Names: Ticilmumab
  Arms: Durvalumab +Tremelimumab + 8 Gy in 1 fraction; Durvalumab +Tremelimumab +5 Gy in 5 fractions; Tremelimumab + 5 Gy in 5 fractions; Tremelimumab + 8 Gy in 1 fraction
Radiation: Sterostatic body radiation therapy (SBRT) — 8 Gray (Gy) x 1; 5Gy x 5
  Other Names: Sterostatic ablative radiotherapy

SUMMARY:
Background:

- Stereotactic body radiation therapy (SBRT) is used to treat cancer. It is a way of giving very focused beams of radiation to tumors. Researchers think that the drugs being used in this study might work better when combined with SBRT in people with pancreatic cancer.

Objective:

- To study the safety and effectiveness of Durvalumab (MEDI4736) and/or tremelimumab with SBRT.

Eligibility:

- People 18 and older who have pancreatic cancer that has not responded or to chemotherapy. They must be candidates for radiation but not resection.

Design:

* Participants will be screened with medical history and physical exam. They will have blood tests. Their tumor will be measured using computerized tomography (CT) or magnetic resonance imaging (MRI).
* Participants will have their tumor biopsied with a needle. They will have also have a biopsy after cycle 1.
* Participants will get 1 or 2 drugs in combination with the SBRT.
* For MEDI4736, the duration of each cycle will be 28-days. Participants will get the drug through an intravenous (IV) infusion twice in each cycle (Days 1 and 15).
* For tremelimumab, the duration of the first 6 cycles will each last 28 days. Then the duration of the last 3 cycles will change to 12 weeks. Participants will get the drug through an IV once in each cycle.
* All participants will have SBRT. Some will get 1 dose of radiation and some will get 5. CT scans will map their tumor.
* Participants will have medical history, physical exam, and blood tests in each cycle. They will have a CT scan or MRI every 8 weeks. Cycles will continue for up to 12 months.
* Participants will be contacted yearly for follow-up.

DETAILED DESCRIPTION:
Background:

Tremelimumab is a monoclonal antibody against cytotoxic T-lymphocyte-associated protein 4 (CTLA4). Anti-CTLA4 therapy has been shown to enhance anti-tumor immunity by blocking tumor-induced immune suppression of cytotoxic T cells.

Durvalumab is a human monoclonal antibody directed against Programmed death-ligand 1 (PD-L1). Blockage of ligation between PD-L1 and Programmed cell death protein 1 (PD1) induces local immune activation and prevent anergy and exhaustion of effectors T-cells.

Several studies have documented an increase in peripheral antitumor immunity following radiation. This effect is evidently too weak to be clinically relevant, but has the potential to be boosted by immune modulation.

The underlying hypothesis of this study is that the effect of Immune Checkpoint inhibitor (Durvalumab with or without Tremelimumab) treatment can be enhanced by radiation in patients with advanced pancreatic carcinoma.

Objective:

To determine the safety, tolerability and feasibility of immune checkpoint inhibition [comprising either Durvalumab alone, or combined Durvalumab and Tremelimumab] in combination with stereotactic body radiation therapy (SBRT) in patients with unresectable pancreatic cancer.

Eligibility:

Histologically confirmed metastatic pancreatic cancer with primary in-situ (or locally-recurrent) with at least 1 measurable metastatic lesion by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria and accessible for biopsy. There is no limit to the number of prior chemotherapy regimens received.

Patients must be greater than or equal to 18 years of age and have a performance status (Eastern Cooperative Oncology Group (ECOG)) less than or equal to 1

Life expectancy of greater than 3 months.

Acceptable organ and bone marrow function.

Patients must not have had standard of care chemotherapy, radiotherapy, or major surgery within the last 2 weeks prior to entering the study. For recent experimental therapies a 28 day period of time must have elapsed before commencing protocol treatment.

No active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease, diverticulitis with the exception of diverticulosis, celiac disease, irritable bowel disease; Wegner syndrome; Hashimoto syndrome; Graves disease; rheumatoid arthritis, hypophysitis, uveitis, etc.) within the past 3 years prior to the start of treatment.

No active or history of inflammatory bowel disease (colitis, Crohn's), irritable bowel disease, celiac disease, or other serious, chronic, gastrointestinal conditions associated with diarrhea. No active or history of systemic lupus erythematosus, Wegeners granulomatosis.

Design:

Subjects will be assigned to 4 arms

Anti-PDL1 (Durvalumab) in combination with radiation (8 Gray (Gy) in fraction)

- Anti-PDL1 (Durvalumab) in combination with radiation (5 Gy in 5 fractions)

Anti-PDL1 (Durvalumab) and anti-CTLA4 (Tremelimumab) in combination with radiation (8 Gy in 1 fractions)

- Anti-PDL1 (Durvalumab) and anti-CTLA4 (Tremelimumab) in combination with radiation (5 Gy in 5 fractions).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histopathological confirmation of pancreatic adenocarcinoma prior to entering this study by the Laboratory of Pathology of the National Cancer Institute (NCI) to entering this study by the Laboratory of Pathology of the NCI prior to entering this study
* Patients must have disease that is not amenable to potentially curative resection. Primary in-situ (or locally-recurrent) tumor must be present and, in the opinion of radiation oncology, be amenable to radiation therapy as planned in the protocol. Each case will be discussed at GI tumor board with multidisciplinary team.
* Patients must have at least 1 measurable metastatic lesion by Response Evaluation in Solid Tumors (RECIST) 1.1 criteria.
* There is no limit to the number of prior chemotherapy regimens received. Patients must have received at least one line of prior systemic chemotherapy for advanced unresectable and/or metastatic disease.
* Age greater than or equal to 18 years
* Life expectancy of greater than 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count - > 1,000/mcL
  * Platelets - greater than or equal to 100,000/mcL
  * total bilirubin - Bili should be less than or equal to 2 x upper limit of normal (ULN) (patients with Gilbert's Syndrome must have a total bilirubin less than 3.0 mg/dL)
  * serum albumin - greater than or equal 2.5 g/dL

Patients are eligible with alanine aminotransferase (ALT) or aspartate aminotransaminase (AST) up to 3 x ULN. (up to 5 x ULN if liver metastases present)

--Creatinine - < 2X institution upper limit of normal

OR

--creatinine clearance - >45 mL/min/1.73 m(2), for patients with creatinine levels above institutional normal

* Patients must have recovered from any acute toxicity related to prior therapy, including surgery. Toxicity should be less than or equal to grade 1 or returned to baseline.
* Patient must be able to understand and willing to sign a written informed consent document.

EXCLUSION CRITERIA:

* Malignant ascites that is clinically detectable by physical examination or is symptomatic. Evidence of radiographic ascites that is not clinically significant will not be an exclusion criterion.
* Any prior Grade greater than or equal to 3 imAE while receiving immunotherapy, including anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA4) treatment, or any unresolved imAE > Grade 1. Note: Active or history of vitiligo will not be a basis for exclusion.
* Patients must not have had standard of care chemotherapy, radiotherapy, or major surgery within the last 2 weeks prior to entering the study. Note: Local surgeries for isolated lesions for palliative intent are acceptable. For recent experimental therapies a 28 day period of time must have elapsed before commencing protocol treatment.
* Patients with known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Uncontrolled intercurrent illness, including, but not limited to, ongoing or active infection, current pneumonitis, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events from Durvalumab (MEDI4736) or tremelimumab, or compromise the ability of the subject to give written informed consent.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease, diverticulitis with the exception of diverticulosis, celiac disease, irritable bowel disease; Wegner syndrome; Hashimoto syndrome; Graves disease; rheumatoid arthritis, hypophysitis, uveitis, etc.) within the past 3 years prior to the start of treatment. The following are exceptions to this criterion:

  * Subjects with vitiligo or alopecia
  * Requirement for intermittent use of bronchodilators or local steroid injections
  * Subjects with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement, or psoriasis not requiring systemic treatment
* History of primary immunodeficiency or history of active tuberculosis. Note: Latent tuberculosis will not be a basis for exclusion.
* Diverticulitis (either active or history of) within the past 2 years. Note that diverticulosis is permitted.
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of Information and Consent and compliance with the requirements of the protocol.
* True positive test results for hepatitis A (Immunoglobulin M (IgM) positive). Subjects with a history of hepatitis A with Immunoglobulin G (IgG) blood test are not excluded. True positive test results hepatitis B, or C infection.
* Active or history of inflammatory bowel disease (colitis, Crohn's), irritable bowel disease, celiac disease, or other serious, chronic, gastrointestinal conditions associated with diarrhea. Active or history of systemic lupus erythematosus or Wegeners granulomatosis.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of MEDI4736 and tremelimumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, and topical steroids
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent
  * Steroids as premedication for hypersensitivity reactions (eg, computed tomography (CT) scan premedication)
* History of sarcoidosis syndrome.
* Patients should not be vaccinated with live attenuated vaccines within 1 month of starting Tremelimumab and MEDI4736 treatment. Subjects, if enrolled, should not receive live vaccine during the study and 180 days after the last dose of both drugs.
* Human immunodeficiency virus (HIV)-positive patients receiving anti-retroviral therapy are excluded from this study due to the possibility of pharmacokinetic interactions between antiretroviral medications and Tremelimumab or MEDI4736. HIV positive patients not receiving antiretroviral therapy are excluded due to the possibility that Tremelimumab or MEDI4736 may worsen their condition and the likelihood that the underlying condition may obscure the attribution of adverse events.
* History of hypersensitivity reaction to human or mouse antibody products.
* Pregnancy and breast feeding are exclusion factors. The effects of Tremelimumab and MEDI4736 on the developing human fetus are unknown. Enrolled patients must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, the duration of study participation and 180 days (female patients) or 90 days (male patients) after the end of the treatment. In addition male patients must refrain from sperm donation for 90 days after the final dose of investigational product. Female patients must refrain from egg cell donation for 180 days after the final dose of investigational product. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim F Greten, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moore MJ, Goldstein D, Hamm J, Figer A, Hecht JR, Gallinger S, Au HJ, Murawa P, Walde D, Wolff RA, Campos D, Lim R, Ding K, Clark G, Voskoglou-Nomikos T, Ptasynski M, Parulekar W; National Cancer Institute of Canada Clinical Trials Group. Erlotinib plus gemcitabine compared with gemcitabine alone in patients with advanced pancreatic cancer: a phase III trial of the National Cancer Institute of Canada Clinical Trials Group. J Clin Oncol. 2007 May 20;25(15):1960-6. doi: 10.1200/JCO.2006.07.9525. Epub 2007 Apr 23. PMID 17452677
- [Background] Reyes-Gibby CC, Chan W, Abbruzzese JL, Xiong HQ, Ho L, Evans DB, Varadhachary G, Bhat S, Wolff RA, Crane C. Patterns of self-reported symptoms in pancreatic cancer patients receiving chemoradiation. J Pain Symptom Manage. 2007 Sep;34(3):244-52. doi: 10.1016/j.jpainsymman.2006.11.007. Epub 2007 May 21. PMID 17513082
- [Background] Moertel CG, Childs DS Jr, Reitemeier RJ, Colby MY Jr, Holbrook MA. Combined 5-fluorouracil and supervoltage radiation therapy of locally unresectable gastrointestinal cancer. Lancet. 1969 Oct 25;2(7626):865-7. doi: 10.1016/s0140-6736(69)92326-5. No abstract available. PMID 4186452
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-C-0027.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Durvalumab + 8 Gray (Gy) in 1 Fraction | Durvalumab +5 Gy in 5 Fractions | Durvalumab +Tremelimumab + 8 Gy in 1 Fraction | Durvalumab +Tremelimumab +5 Gy in 5 Fractions
Started | 14 | 11 | 19 | 21
Received Radiation Therapy Only | 0 | 1 | 1 | 1
Completed | 14 | 10 | 19 | 20
Not Completed | 0 | 1 | 0 | 1
Not completed — Did not receive treatment | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Durvalumab + 8 Gray (Gy) in 1 Fraction | Durvalumab +5 Gy in 5 Fractions | Durvalumab +Tremelimumab + 8 Gy in 1 Fraction | Durvalumab +Tremelimumab +5 Gy in 5 Fractions | Total
Number analyzed (Participants) | 14 | 11 | 19 | 21 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 6 | 13 | 12 | 41
  >=65 years | 4 | 5 | 6 | 9 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.75 (9.27) | 61.70 (6.36) | 64.26 (11.77) | 65.31 (9.58) | 63.26 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 9 | 4 | 25
  Male | 7 | 6 | 10 | 17 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 14 | 11 | 18 | 21 | 64
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 3 | 4 | 8
  White | 11 | 11 | 16 | 17 | 55
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 11 | 19 | 21 | 65

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events in Each Cohort With Grade 1 Through 5 Related to Study Drug
Description: Adverse Events (AEs) are reported by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Grade 1=Mild, Grade 2= Moderate, Grade 3 = Severe, Grade 4 = Life-threatening, and Grade 5 = Fatal.
Time Frame: Participants were assessed from the start of study treatment at Cycle 1 then after every cycle (1 cycle = 28 days) of protocol treatment until 30 days after they were taken off treatment, approximately 4.0 months.
Measure: Number; unit: Adverse events
Groups:
- Cohort A Dose Level A1: Durvalumab + 8 Gray (Gy) in 1 fraction
  Durvalumab: 10 mg/kg, mg intravenous (IV), every two weeks, or 1500 mg, IV, every four weeks.
  Sterostatic body radiation therapy (SBRT): 8 Gray (Gy) x 1; 5Gy x 5
- Cohort A Dose Level A2: Durvalumab +5 Gy in 5 fractions
  Durvalumab: 10 mg/kg, mg intravenous (IV), every two weeks, or 1500 mg, IV, every four weeks.
  Sterostatic body radiation therapy (SBRT): 8 Gray (Gy) x 1; 5Gy x 5
- Cohort C Dose Level C1: Durvalumab +Tremelimumab + 8 Gy in 1 fraction
  Durvalumab: 10 mg/kg, mg intravenous (IV), every two weeks, or 1500 mg, IV, every four weeks.
  Tremelimumab: 75 mg IV, every 4 weeks for 16 weeks
  Sterostatic body radiation therapy (SBRT): 8 Gray (Gy) x 1; 5Gy x 5
- Cohort C Dose Level C2: Durvalumab +Tremelimumab +5 Gy in 5 fractions
  Durvalumab: 10 mg/kg, mg intravenous (IV), every two weeks, or 1500 mg, IV, every four weeks.
  Tremelimumab: 75 mg IV, every 4 weeks for 16 weeks
  Sterostatic body radiation therapy (SBRT): 8 Gray (Gy) x 1; 5Gy x 5
Arm/Group | Cohort A Dose Level A1 | Cohort A Dose Level A2 | Cohort C Dose Level C1 | Cohort C Dose Level C2
Number analyzed (Participants) | 14 | 10 | 19 | 20
Adverse events
  Grade 1 Abdominal pain | 0 | 0 | 0 | 1
  Grade 1 Alanine aminotransferase increased | 1 | 0 | 0 | 5
  Grade 1 Alkaline Phosphatase increased | 0 | 2 | 0 | 2
  Grade 1 Anemia | 3 | 3 | 9 | 9
  Grade 1 Anorexia | 1 | 0 | 0 | 3
  Grade 1 Atrial fibrillation | 0 | 0 | 0 | 1
  Grade 1 Aspartate aminotransferase increased | 1 | 0 | 1 | 6
  Grade 1 Back pain | 0 | 0 | 0 | 1
  Grade 1 Blood bilirubin increased | 0 | 0 | 1 | 1
  Grade 1 Cough | 0 | 0 | 0 | 1
  Grade 1 Creatinine increased | 0 | 0 | 0 | 1
  Grade 1 Diarrhea | 0 | 1 | 1 | 7
  Grade 1 Dizziness | 0 | 0 | 0 | 1
  Grade 1 Dry mouth | 1 | 0 | 0 | 0
  Grade 1 Dysgeusia | 0 | 0 | 1 | 0
  Grade 1 Endocrine disorders,Other, Elevated T3, T4 | 0 | 0 | 1 | 0
  Grade 1 Eye disorders - decr. in near vision,bilat | 0 | 1 | 0 | 0
  Grade 1 - Fatigue | 1 | 2 | 0 | 7
  Grade 1 Fever | 1 | 1 | 1 | 1
  Grade 1 Headache | 0 | 2 | 0 | 0
  Grade 1 Hemorrhoidal hemorrhage | 1 | 0 | 0 | 0
  Grade 1 Hoarseness | 0 | 0 | 1 | 0
  Grade 1 Hyperglycemia | 0 | 0 | 2 | 0
  Grade 1 - Hyperkalemia | 0 | 0 | 0 | 1
  Grade 1 Hyperuricemia | 0 | 0 | 0 | 1
  Grade 1 Hypoalbuminemia | 0 | 0 | 0 | 5
  Grade 1 Hypocalcemia | 0 | 0 | 0 | 1
  Grade 1 - Hyponatremia | 2 | 0 | 3 | 4
  Grade 1 Hypothyroidism | 0 | 0 | 0 | 1
  Grade 1 Infusion related reaction | 0 | 0 | 0 | 2
  Grade 1 Lymphocyte count decreased | 15 | 20 | 17 | 26
  Grade 1 Mucositis | 0 | 0 | 0 | 1
  Grade 1 Musculoskeletal & connective tissue | 0 | 3 | 0 | 0
  Grade 1 Nausea | 0 | 1 | 3 | 2
  Grade 1 Neutrophil count decreased | 0 | 0 | 0 | 1
  Grade 1 Pain | 0 | 0 | 0 | 1
  Grade 1 Platelet count decreased | 2 | 0 | 7 | 13
  Grade 1 Pruritis | 1 | 1 | 2 | 3
  Grade 1 Rash maculo-papular | 0 | 1 | 1 | 2
  Grade 1 Serum amylase increased | 0 | 0 | 0 | 3
  Grade 1 - Skin/subc tissue disorder - Night sweats | 0 | 0 | 1 | 1
  Grade 1 Skin/subc tissue disorder - Rash | 0 | 0 | 1 | 0
  Grade 1 Skin/subc tissue - Psoriasis | 0 | 1 | 0 | 0
  Grade 1 Skin/subc tissue disorder - Itching | 0 | 1 | 1 | 0
  Grade 1 Skin/subc tissue disorder-Skinpeeling hand | 0 | 0 | 1 | 0
  Grade 1 Vertigo | 0 | 1 | 0 | 0
  Grade 1 Vomiting | 0 | 0 | 1 | 4
  Grade 1 Weight loss | 0 | 0 | 0 | 1
  Grade 1 White blood cell decreased | 1 | 4 | 1 | 7
  Grade 2 Abdominal pain | 0 | 0 | 0 | 1
  Grade 2 Anemia | 3 | 1 | 9 | 10
  Grade 2 Anorexia | 0 | 0 | 0 | 2
  Grade 2 Autoimmune disorder | 0 | 0 | 0 | 1
  Grade 2 Diarrhea | 0 | 1 | 2 | 4
  Grade 2 Dysgeusia | 0 | 0 | 0 | 1
  Grade 2 Endocrine disorders - TSH elev-Hypothyroid | 0 | 0 | 1 | 0
  Grade 2 Fatigue | 0 | 0 | 2 | 5
  Grade 2 Fecal incontinence | 0 | 1 | 0 | 0
  Grade 2 Fever | 0 | 0 | 0 | 1
  Grade 2 Gastroesophageal reflux disease | 0 | 1 | 0 | 0
  Grade 2 Hyperglycemia | 0 | 0 | 1 | 0
  Grade 2 Hypoalbuminemia | 0 | 0 | 0 | 1
  Grade 2 Hypothyroidism | 0 | 0 | 1 | 0
  Grade 2 Hypophosphatemia | 1 | 0 | 0 | 0
  Grade 2 Infusion related reaction | 0 | 0 | 1 | 0
  Grade 2 Lymphocyte count decreased | 7 | 19 | 15 | 30
  Grade 2 Malaise | 0 | 0 | 0 | 2
  Grade 2 Nausea | 0 | 0 | 0 | 3
  Grade 2 Neutrophil count decreased | 0 | 0 | 2 | 1
  Grade 2 Platelet count decreased | 0 | 0 | 1 | 2
  Grade 2 Rash maculo-papular | 0 | 0 | 0 | 1
  Grade 2 Weight loss | 0 | 0 | 0 | 2
  Grade 2 White blood cell count | 0 | 2 | 1 | 0
  Grade 3 Anemia | 0 | 0 | 2 | 3
  Grade 3 Anorexia | 0 | 0 | 0 | 1
  Grade 3 Colitis | 0 | 0 | 0 | 2
  Grade 3 Dehydration | 0 | 0 | 0 | 3
  Grade 3 Diarrhea | 0 | 0 | 0 | 3
  Grade 3 Fatigue | 0 | 0 | 1 | 1
  Grade 3 Hyperthyroidism | 0 | 0 | 0 | 1
  Grade 3 Lymphocyte count decreased | 3 | 7 | 6 | 18
  Grade 3 Nausea | 0 | 0 | 0 | 2
  Grade 3 Serum amylase increased | 0 | 0 | 1 | 0
  Grade 3 Vomiting | 0 | 0 | 0 | 2
  Grade 4 Lymphocyte count decreased | 0 | 0 | 2 | 2

2. Secondary Outcome: Plasma Pharmacokinetic (PK)
Description: Drug level in blood
Time Frame: 30 days after treatment
Population: The pharmacokinetic studies were not done since the company were not interested in this after the samples were collected
Arm/Group | Cohort A Dose Level A1 | Cohort A Dose Level A2 | Cohort C Dose Level C1 | Cohort C Dose Level C2
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants With 6-month Overall Survival
Description: Participants who survived at least 6 months after therapy.
Time Frame: 6 month
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A Dose Level A1 | Cohort A Dose Level A2 | Cohort C Dose Level C1 | Cohort C Dose Level C2
Number analyzed (Participants) | 14 | 10 | 19 | 20
percentage of participants | 26 | 58 | 12 | 40

4. Secondary Outcome: Overall Survival
Description: Amount of time participants survived after therapy.
Time Frame: From study entry to death or date of last contact, whichever occurs first, up to 2 years of follow-up
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A Dose Level A1 | Cohort A Dose Level A2 | Cohort C Dose Level C1 | Cohort C Dose Level C2
Number analyzed (Participants) | 14 | 10 | 19 | 20
Months | 3.3 [1.2 to 6.6] | 9.0 [0.5 to 18.4] | 2.1 [1.1 to 4.3] | 4.2 [2.9 to 9.3]

5. Secondary Outcome: Tumor Response Assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as Measured by Computed Tomography (CT) and Magnetic Resonance Imaging (MRI)
Description: Progressive disease (PD): >=20% increase in sum of longest diameter (LD) of target lesion(s), taking as reference smallest sum LD recorded since treatment started. Complete response (CR): disappearance of all target lesions. Partial response (PR): >=30% decrease in sum of LD of target lesion(s), taking as reference baseline sum LD. Stable disease (SD): neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD.
Time Frame: At screening then every 8 weeks until disease progression or patient is taken off the trial, whichever comes first, approximately 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A Dose Level A1 | Cohort A Dose Level A2 | Cohort C Dose Level C1 | Cohort C Dose Level C2
Number analyzed (Participants) | 14 | 10 | 19 | 20
Participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 1 | 0 | 0 | 1
  Stable Disease | 3 | 4 | 2 | 5
  Progressive Disease | 4 | 4 | 6 | 10

6. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is the defined as the median amount of time subject survives without disease progression after treatment. Progression is assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) and is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). NOTE: While RECIST Progressive Disease (PD) will be noted and recorded the immune-related (IR) RECIST criteria will be applied to determine discontinuation of study treatment. For modified Immune-Related Response Criteria (irRC), only target and measurable lesions are taken into account.
Time Frame: From study entry to disease progression, death or date of last contact, whichever occurs first, an average of 6 months
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A Dose Level A1 | Cohort A Dose Level A2 | Cohort C Dose Level C1 | Cohort C Dose Level C2
Number analyzed (Participants) | 14 | 10 | 19 | 20
Months | 1.7 [0.8 to 2.0] | 2.5 [0.1 to 3.7] | 0.9 [0.7 to 2.1] | 2.3 [1.9 to 3.4]

7. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 18 months and 4 days for Cohort 1/Dose Level A1, 23 months and 29 days for Cohort 2/Dose Level A2, 32 months and 19 days for Cohort C/Dose Level C1, and 44 months and 18 days for Cohort C/Dose
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab + 8 Gray (Gy) in 1 Fraction | Durvalumab +5 Gy in 5 Fractions | Durvalumab +Tremelimumab + 8 Gy in 1 Fraction | Durvalumab +Tremelimumab +5 Gy in 5 Fractions
Number analyzed (Participants) | 14 | 11 | 19 | 20
Participants | 14 | 10 | 19 | 20

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 18 months and 4 days for Cohort 1/Dose Level A1, 23 months and 29 days for Cohort 2/Dose Level A2, 32 months and 19 days for Cohort C/Dose Level C1, and 44 months and 18 days for Cohort C/Dose Level C2.
Description: One patient did not get treated in Cohort 2/Dose Level A2 and Cohort C/Dose Level C2.
Arm/Group | Durvalumab + 8 Gray (Gy) in 1 Fraction | Durvalumab +5 Gy in 5 Fractions | Durvalumab +Tremelimumab + 8 Gy in 1 Fraction | Durvalumab +Tremelimumab +5 Gy in 5 Fractions
All-Cause Mortality (participants affected / at risk) | 14/14 | 8/11 | 2/19 | 3/20
Serious Adverse Events (participants affected / at risk) | 6/14 | 2/11 | 11/19 | 12/20
Other Adverse Events (participants affected / at risk) | 14/14 | 10/11 | 19/19 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab + 8 Gray (Gy) in 1 Fraction (N=14) | Durvalumab +5 Gy in 5 Fractions (N=11) | Durvalumab +Tremelimumab + 8 Gy in 1 Fraction (N=19) | Durvalumab +Tremelimumab +5 Gy in 5 Fractions (N=20)
Death NOS (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (4) | 7 (8)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac disorders - Other, pulm embolism (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain - cardiac (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, Abdominal cramping (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Endocarditis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Gastrointestinal disorders - Other, Liver abscess (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Ileal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Infections and infestations - Other, pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab + 8 Gray (Gy) in 1 Fraction (N=14) | Durvalumab +5 Gy in 5 Fractions (N=11) | Durvalumab +Tremelimumab + 8 Gy in 1 Fraction (N=19) | Durvalumab +Tremelimumab +5 Gy in 5 Fractions (N=20)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Edema trunk (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Gastrointestinal disorders - Other,bile duct obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 2 (3) | 3 (3) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 5 (5) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Eye disorders - Other - decrease in near vision bilat eye, blurry vision
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Infections and infestations - Other, Strep and haemophilus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Muscular other: Bilateral leg cramps
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Nervous system disorders - Other, specify: Restless leg syndrome symptoms
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Psychiatric disorders - Other: Fogginess
Rectal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Retinal vascular disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight gain (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Investigations) | 8 (10) | 1 (1) | 7 (9) | 9 (17)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood and lymphatic system disorders - Other, Increased PT (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endocrine disorders - Other, Elevated T3, T4 (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 7 (17) | 9 (15) | 6 (13) | 10 (30)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 3 (3) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Respiratory, thoracic and mediastinal disorders - Other: pneumonia
Serum amylase increased (Investigations) | 1 (2) | 2 (2) | 3 (3) | 2 (9)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (3)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4) | 6 (7) | 6 (7)
Weight loss (Investigations) | 1 (1) | 2 (2) | 3 (3) | 6 (7)
White blood cell decreased (Investigations) | 4 (11) | 5 (16) | 2 (10) | 5 (13)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (5) | 4 (10) | 5 (11) | 12 (25)
Activated partial thromboplastin time prolonged (Investigations) | 10 (23) | 6 (19) | 3 (5) | 8 (10)
Alanine aminotransferase increased (Investigations) | 6 (15) | 2 (2) | 6 (7) | 11 (30)
Alkaline phosphatase increased (Investigations) | 9 (24) | 5 (9) | 9 (15) | 18 (43)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 10 (28) | 9 (30) | 15 (37) | 16 (46)
Ascites (Gastrointestinal disorders) | 3 (3) | 0 (0) | 7 (7) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 7 (15) | 3 (6) | 9 (13) | 12 (25)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Autoimmune disorder (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (7) | 2 (2) | 6 (10)
Bloating (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (2) | 2 (2)
Blood bilirubin increased (Investigations) | 6 (14) | 2 (2) | 6 (10) | 5 (15)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (5) | 5 (9) | 4 (4) | 8 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 3 (3) | 3 (4)
Creatinine increased (Investigations) | 3 (6) | 1 (1) | 1 (1) | 3 (5)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 5 (9) | 8 (9) | 8 (19)
Dizziness (Nervous system disorders) | 2 (2) | 5 (7) | 2 (2) | 6 (7)
Dysgeusia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 4 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (3) | 4 (5) | 6 (7)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 2 (3) | 3 (6) | 4 (5) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 7 (9) | 8 (10) | 7 (9) | 15 (22)
Fever (General disorders) | 4 (5) | 3 (4) | 3 (3) | 5 (11)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Generalized muscle weakness (General disorders) | 2 (4) | 1 (1) | 2 (4) | 3 (3)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 2 (3) | 1 (1) | 4 (4)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (7) | 0 (0) | 5 (11) | 4 (11)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 3 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 3 (5)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (5) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (3) | 4 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 (24) | 8 (19) | 13 (31) | 16 (37)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (4) | 3 (3) | 4 (9) | 4 (6)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hypokalemia (Metabolism and nutrition disorders) | 6 (18) | 3 (6) | 1 (1) | 8 (11)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (8) | 2 (2) | 5 (6) | 5 (10)
Hyponatremia (Metabolism and nutrition disorders) | 10 (22) | 3 (8) | 11 (22) | 9 (24)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (12) | 1 (1) | 8 (12) | 7 (12)
Hypotension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 3 (3)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (3) | 2 (2) | 4 (4)
Lethargy (General disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 12 (44) | 10 (54) | 16 (52) | 18 (92)
Malaise (General disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (6) | 3 (5) | 9 (12) | 7 (9)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (4) | 2 (2) | 1 (4)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 8 (14) | 4 (8) | 2 (3) | 5 (6)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 7 (17) | 8 (13) | 5 (13) | 12 (32)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, weakness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, Fullness/Bloating (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Gastrointestinal disorders - Other: cramping pain, muscle spasm
Gastrointestinal disorders - Other, Specify (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Gastrointestinal disorders - Other: muscle spasm
Gastrointestinal disorders - Other, Abdominal cramping (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Gastrointestinal disorders - Other: cramping
Gastrointestinal disorders - Other, Upper abdominal soreness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Gastrointestinal disorders - Other: greasiness to stool
Infections and infestations - Other, C-diff. infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, yeast infection - rectal area (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — infections and infestations - Other: portacath
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Musculoskeletal and connective tissue disorder - Other, Upper back pain
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) — Musculoskeletal and connective tissue disorder - Other: cramping in balls of feet bilaterally
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Skin and subcutaneous tissue disorders -Other: itching
Skin and subcutaneous tissue disorders -Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Skin and subcutaneous tissue disorders -Other: palpable mass
Endocrine disorders - Other, TSH elevated - hypothyroidsim (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders -Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Skin and subcutaneous tissue disorders -Other: other night sweats
Skin and subcutaneous tissue disorders -Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Skin and subcutaneous tissue disorders -Other: itching
Skin and subcutaneous tissue disorders -Other, mouth sore (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders -Other, Skin peeling - hand (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders -Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Skin and subcutaneous tissue disorders -Other: hives
Skin and subcutaneous tissue disorders -Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Skin and subcutaneous tissue disorders -Other: rash

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2018-08-24): https://cdn.clinicaltrials.gov/large-docs/61/NCT02311361/Prot_SAP_000.pdf
  • Informed Consent Form: Arms A1 and A2 Consent (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/61/NCT02311361/ICF_001.pdf
  • Informed Consent Form: Arms C1 and C2 Consent (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/61/NCT02311361/ICF_002.pdf